CLINICAL TRIAL: NCT07298057
Title: Effectiveness of Scaling and Root Planing With and Without Minocycline Microspheres (Arestin) in Improving Periodontal and Glycemic Outcomes in Diabetic Patients With Periodontitis: A Randomized Controlled Trial
Brief Title: Effect of Arestin-Enhanced SRP on Periodontal and Glycemic Outcomes in Diabetics
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: OraPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY20250753
Record Dates: First submitted 2025-12-11; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis, Diabetes Mellitus Type 2
Keywords: Scaling and Root Planing; Arestin; Diabetes Mellitus Type 2
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus, Type 2; cyclopia sequence | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental): Minocycline microspheres (Arestin®) / (4 mg per cartridge) prefilled delivery syringe / Arestin will be placed in the pocket only one time after scaling and root planing.
  Interventions: Drug: local antibiotic application of topical minocycline
- Control Group (Active Comparator): Scaling and Root Planing Alone
  Interventions: Procedure: Scaling and Root Planing

INTERVENTIONS:
Drug: local antibiotic application of topical minocycline — Scaling and Root planing + local application of Arestin ( Minocycline microsphere)
  Other Names: Arestin Minocicline microsphere
  Arms: Test Group
Procedure: Scaling and Root Planing — Only scaling and root planing
  Arms: Control Group

SUMMARY:
Periodontitis is a prevalent chronic inflammatory disease that exacerbates systemic inflammation and poses challenges for glycemic control in diabetic patients. While scaling and root planing (SRP) remains the cornerstone of periodontal therapy, adjunctive treatments such as Arestin (minocycline microspheres) have shown promise in enhancing clinical outcomes. This study aims to evaluate the impact of adding Arestin to SRP on periodontal pocket closure, glycemic control, and systemic inflammation in diabetic patients with periodontitis.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years) with type 2 diabetes mellitus (HbA1c ≥ 7.0% and ≤9.5%)
2. Diagnosed with moderate to severe periodontitis (≥5 mm probing pocket depth in at least 6 distinct interproximal sites, on different teeth)
3. At least 16 teeth present
4. No periodontal treatment in the last 6 months

Exclusion Criteria:

1. Allergy to minocycline or tetracycline
2. Unable to receive or to tolerate local anesthesia
3. Unable to tolerate tooth instrumentation with ultrasonic instruments.
4. Require IV sedation to receive scaling and root planing
5. Use of antibiotics within the past 3 months
6. Pregnancy or breastfeeding
7. Morbid Obesity (BMI 40+)
8. Smokers or patients with poorly controlled systemic diseases other than diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Pocket Closure | Baseline, 3 Months, 6 Months
  Pocket Depth (PD ≤4 mm)

SECONDARY OUTCOMES:
Changes in Glycemic Control (HbA1c) | Baseline, 3 Months, 6 Months
  Changes in Blood Sugar Level
Changes in C-reactive Protein Level (CRP) | Baseline, 3 Months, 6 Months
  Changes in Systemic Inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Gian Pietro Schincaglia, DDS, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared with other researchers. Only de-identified, cumulative data (summary-level results) will be shared with the study sponsor (OraPharma) after study completion. No identifiable participant information such as name, date of birth, or contact details will be disclosed. All collected data will remain securely stored within Case Western Reserve University and will only be accessed by the study investigators and authorized university or regulatory personnel.

REFERENCES:
- [Result] Skaleric U, Schara R, Medvescek M, Hanlon A, Doherty F, Lessem J. Periodontal treatment by Arestin and its effects on glycemic control in type 1 diabetes patients. J Int Acad Periodontol. 2004 Oct;6(4 Suppl):160-5. PMID 15536785
- [Result] Simpson TC, Clarkson JE, Worthington HV, MacDonald L, Weldon JC, Needleman I, Iheozor-Ejiofor Z, Wild SH, Qureshi A, Walker A, Patel VA, Boyers D, Twigg J. Treatment of periodontitis for glycaemic control in people with diabetes mellitus. Cochrane Database Syst Rev. 2022 Apr 14;4(4):CD004714. doi: 10.1002/14651858.CD004714.pub4. PMID 35420698
- [Result] Preshaw PM, Alba AL, Herrera D, Jepsen S, Konstantinidis A, Makrilakis K, Taylor R. Periodontitis and diabetes: a two-way relationship. Diabetologia. 2012 Jan;55(1):21-31. doi: 10.1007/s00125-011-2342-y. Epub 2011 Nov 6. PMID 22057194